CLINICAL TRIAL: NCT02868242
Title: A Phase 2, Open-label Study to Investigate the Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed Dose Combination in the Treatment of Hepatitis C Virus (HCV) Infection in Pediatric Subjects Undergoing Cancer Chemotherapy
Brief Title: Efficacy and Safety of Ledipasvir/Sofosbuvir Fixed Dose Combination in the Treatment of Hepatitis C Virus (HCV) Infection in Pediatric Participants Undergoing Cancer Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-1904
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV genotype 1 or 4 (GT-1 or GT-4); Direct Acting Antiviral; Combination Therapy; Hepatitis C, Chronic; Liver Diseases; Virus Diseases
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Virus Diseases | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LDV/SOF (Experimental): Participants will receive LDV/SOF 90/400 mg fixed dose combination (FDC) (1x 90/400 mg tablet or 4 x 22.5/100 mg tablets based on swallowability assessment during screening) for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — Tablet(s) administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) in treating hepatitis C virus (HCV) infection in pediatric participants who are undergoing cancer chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 12 to <18 years
* Parent or legal guardian must provide written informed consent
* Treatment naïve or experienced children with genotype 1 or 4 HCV infection, and are on a maintenance cancer chemotherapy regimen
* Receiving a protocol-approved maintenance chemotherapy regimen for a hematological malignancy
* Chronic HCV infection (≥ 6 months) documented by medical history or liver biopsy
* Screening laboratory values within defined thresholds
* No History of solid organ or bone marrow transplantation
* No history of clinical hepatic decompensation (eg, ascites, jaundice, encephalopathy, variceal hemorrhage)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- National Cancer Institute, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] El-Sayed MH, Ebeid FSE, Zekri AR, Massetto B, Kersey K, Zhang F, Gaggar A, Elsayed W, El-Haddad A. Ledipasvir-sofosbuvir in Adolescents With Chronic Hepatitis C and Hematological Malignancies Undergoing Chemotherapy. J Pediatr Gastroenterol Nutr. 2022 May 1;74(5):626-630. doi: 10.1097/MPG.0000000000003406. Epub 2022 Feb 10. PMID 35149641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one study site in Egypt. The first participant was screened on 28 August 2016. The last study visit occurred on 03 February 2019.
Pre-assignment Details: 24 participants were screened.
Groups:
- LDV/SOF: LDV/SOF 90/400 mg fixed dose combination (FDC) orally once daily for 12 weeks
Period: Overall Study
Arm/Group | LDV/SOF
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who took at least 1 dose of study drug.
Groups:
- LDV/SOF: LDV/SOF 90/400 mg FDC orally once daily for 12 weeks
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
IL28B [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 6
    CT | 12
    TT | 1
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.3 (1.65)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 12
  ≥ 800,000 IU/mL | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 50 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants | 100.0 [82.4 to 100.0]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event
Time Frame: First dose date up to Week 12
Population: Safety Analysis Set included participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF: LDV/SOF 90/400 mg FDC once daily for 12 weeks
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants | 100.0 [82.4 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants | 100.0 [82.4 to 100.0]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Treatment
Time Frame: Weeks 1, 4, 8, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- LDV/SOF: LDV/SOF FDC 90/400 mg orally once daily for 12 weeks
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants
  Week 1 | 89.5 [66.9 to 98.7]
  Week 4 | 100.0 [82.4 to 100.0]
  Week 8 | 94.7 [74.0 to 99.9]
  Week 12 | 100.0 [82.4 to 100.0]

6. Secondary Outcome: HCV RNA Change From Baseline/Day 1
Time Frame: Baseline; Weeks 1, 4, 8, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
log10 IU/mL
  Change at Week 1 | -3.34 (1.730)
  Change at Week 4 | -3.62 (1.653)
  Change at Week 8 | -3.36 (1.526)
  Change at Week 12 | -3.62 (1.653)

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF
Number analyzed (Participants) | 19
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Week 12 plus 30 days; All-Cause Mortality: First dose date up to Posttreatment Week 24
Description: Safety Analysis Set included participants who took at least 1 dose of study drug.
Arm/Group | LDV/SOF
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=19)
Diarrhoea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=19)
Anaemia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Lip ulceration (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Tongue ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 5
Conjunctivitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 2
Hypophagia (Metabolism and nutrition disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT02868242/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02868242/SAP_001.pdf